CLINICAL TRIAL: NCT03507738
Title: A Phase 1, Randomized, Placebo-controlled, Descending Age, Dose-escalation Study to Assess the Safety and Immunogenicity of an Investigational Non-Replicating Rotavirus Vaccine (MT-5625) in Healthy Adults, Toddlers and Infants
Brief Title: Safety and Immunogenicity of MT-5625 in Healthy Adults, Toddlers and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MT-5625-01
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — RIX4414 vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Adult MT-5625 middle dose (Experimental): Adult receiving intramuscular injection with either middle dose of MT-5625 or placebo
  Interventions: Biological: MT-5625 middle dose; Biological: Placebo
- Adult MT-5625 high dose (Experimental): Adult receiving intramuscular injection with either high dose of MT-5625 or placebo
  Interventions: Biological: MT-5625 high dose; Biological: Placebo
- Toddler MT-5625 middle dose (Experimental): Toddler receiving intramuscular injection with either middle dose of MT-5625 or placebo
  Interventions: Biological: MT-5625 middle dose; Biological: Placebo
- Toddler MT-5625 high dose (Experimental): Toddler receiving intramuscular injection with either high dose of MT-5625 or placebo
  Interventions: Biological: MT-5625 high dose; Biological: Placebo
- Infant MT-5625 low dose (Experimental): Infant receiving intramuscular injection with either low dose of MT-5625 or placebo
  Interventions: Biological: MT-5625 low dose; Biological: Placebo
- Infant MT-5625 middle dose (Experimental): Infant receiving intramuscular injection with either middle dose of MT-5625 or placebo
  Interventions: Biological: MT-5625 middle dose; Biological: Placebo
- Infant MT-5625 high dose (Experimental): Infant receiving intramuscular injection with either high dose of MT-5625 or placebo
  Interventions: Biological: MT-5625 high dose; Biological: Placebo
- Rotarix (Active Comparator): Infant receiving oral administration with Rotarix
  Interventions: Biological: Rotarix

INTERVENTIONS:
Biological: MT-5625 low dose — Intramuscular injection
  Arms: Infant MT-5625 low dose
Biological: MT-5625 middle dose — Intramuscular injection
  Arms: Adult MT-5625 middle dose; Infant MT-5625 middle dose; Toddler MT-5625 middle dose
Biological: MT-5625 high dose — Intramuscular injection
  Arms: Adult MT-5625 high dose; Infant MT-5625 high dose; Toddler MT-5625 high dose
Biological: Rotarix — Oral administration
  Arms: Rotarix
Biological: Placebo — Intramuscular injection
  Arms: Adult MT-5625 high dose; Adult MT-5625 middle dose; Infant MT-5625 high dose; Infant MT-5625 low dose; Infant MT-5625 middle dose; Toddler MT-5625 high dose; Toddler MT-5625 middle dose

SUMMARY:
A study to investigate the safety and reactogenicity of MT-5625 independently in adults aged 18-35 years, toddlers ages 12-24 months, and infants aged 6-10 weeks

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults/toddlers/infants as established by medical history and clinical examination before entering the study
* Adults aged >18 and < 35, toddlers aged >12 and < 24 months, and infants aged > 6 and < 10 weeks at the time of enrollment
* Subject (or Parent/Legal Guardian) willing and able to give written informed consent after the nature of the study has been explained
* Subject (or Parent/Legal Guardian) willing to comply with the study restrictions and study schedule and to remain in the area for the study duration
* Females of potential childbearing must not be pregnant or breastfeeding and willing to use adequate method of contraception during the trial

Exclusion Criteria:

ALL SUBJECTS

* Presence of fever or other acute illness
* Concurrent participation in another clinical trial or receipt of an investigational product during the 30 days prior to randomization
* Suspected or known impairment of immune function
* Known sensitivity to any components of the study vaccine
* History of anaphylactic reaction
* Receipt of immunoglobulin therapy or blood products in last 6 months
* History of chronic immunosuppressive medications (with the exception of inhaled or topical steroids)
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study

ADULTS ONLY

* Have received any vaccine within 4 weeks prior to randomization
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product (IP)
* Any clinically significant abnormalities on 12-lead ECG as judged by the Investigator
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody
* Have any contraindications to parenteral injections ( eg history of bleeding disorder)
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the Investigator
* Donated blood within the 4 weeks prior to randomization

TODDLERS and INFANTS

* Received any vaccine within 14 days of randomization
* Presence of malnutrition or other systemic disorders
* History of congenital abdominal disorders, intussusception or abdominal surgery
* Major congenital or genetic defect

TODDLERS ONLY

* Any positive result on screening for serum hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

INFANTS ONLY

* Infants with history of premature birth (<37 weeks gestational age)
* Infants who have received rotavirus vaccine in the past
* Known sensitivity to any components of the study vaccine, including Rotarix®
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis B core antibody, and hepatitis C antibody
* HIV infection assessed by PCR if mother is not known to be negative (negative test result between 24 weeks gestation and screening).

Ages: 6 Weeks to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with local reactions and reactogenicity events. | Within 7 days after each vaccination
Proportion of subjects reporting adverse events. | Within 28 days after each vaccination

SECONDARY OUTCOMES:
Proportion of subjects with anti-MT-5625 IgG seroresponses | Day 28 after each vaccination
Proportion of subjects with neutralizing antibody responses | Day 28 after each vaccination
Anti-MT-5625 IgG geometric mean titers (GMTs) 28 days after each injection in adults, toddlers, and infants. | Day 28 after each vaccination
Neutralizing antibody GMTs against rotavirus 28 days after each injection in adults, toddlers and infants. | Day 28 after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (2):
- Investigational center, Adelaide, Australia
- Investigational center, Johannesburg, South Africa

REFERENCES:
- [Derived] Kurokawa N, Robinson MK, Bernard C, Kawaguchi Y, Koujin Y, Koen A, Madhi S, Polasek TM, McNeal M, Dargis M, Couture MM, Trepanier S, Forrest BD, Tsutsui N. Safety and immunogenicity of a plant-derived rotavirus-like particle vaccine in adults, toddlers and infants. Vaccine. 2021 Sep 15;39(39):5513-5523. doi: 10.1016/j.vaccine.2021.08.052. Epub 2021 Aug 25. PMID 34454786